CLINICAL TRIAL: NCT05969938
Title: Predicting the Efficacy and Prognosis of Rectal Cancer Patients Receiving Neoadjuvant Chemoradiotherapy Based on Circulating Tumor DNA-minimal Residual Disease Technology : A Prospective, Observational Study
Brief Title: Predicting the Efficacy and Prognosis of Rectal Cancer Patients Based on ctDNA-MRD Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: WeiWei Xiao (Other)
Collaborators: Haplox Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, WeiWei Xiao, Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: B2023-239-01
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Rectal Adenocarcinoma; Circulating Tumor DNA; Minimal Residual Disease; Neoadjuvant Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples including two kinds :1.We will collect tumor tissue samples for WES detection and customized panel.2. We will collect peripheral blood samples for MRD detection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: A total of 50 patients with stage II-III rectal cancer who plan to receive neoadjuvant chemoradiotherapy between the ages of 18-75 years old, and these patients have no distant metastasis, normal main organ function, and can receive long-term follow-up. simultaneously, these patients are required to provide sufficient ' colonoscopy collection ' tumor tissue samples for MRD customization, and sufficient whole blood samples are required for baseline MRD detection.
  Interventions: Diagnostic Test: MRD detection

INTERVENTIONS:
Diagnostic Test: MRD detection — Peripheral blood samples were collected for MRD detection before neoadjuvant chemoradiotherapy, during neoadjuvant chemoradiotherapy, and 3-4 weeks after radical surgery. For patients who achieved cCR after neoadjuvant therapy and adopted the W & W strategy, the sampling time point was 3 months after the start of watching and waiting.

SUMMARY:
The purpose of this study is to study the performance of MRD monitoring in predicting the efficacy and prognosis of neoadjuvant therapy in patients with rectal cancer, and to explore the value of MRD detection in evaluating the prognosis of patients. In this prospective study, 50 patients with stage II-III rectal cancer who are planing to receive neoadjuvant chemoradiotherapy will be enrolled. The tumor tissue will be collected by colonoscopy before treatment and blood samples will be collected before treatment and during treatment.The whole blood samples will receive MRD detection. The change rate and clearance rate of MRD during treatment will be calculated, and will be associated with imaging efficacy evaluation, pathological efficacy evaluation,and prognosis, to determine the performance of MRD in predicting and judging the efficacy of neoadjuvant chemoradiotherapy and postoperative recurrence of rectal cancer.

DETAILED DESCRIPTION:
This study is a prospective, observational study. It is expected to enroll 50 patients with newly diagnosed stage II-III rectal cancer.Before neoadjuvant chemoradiotherapy, tumor tissue will be collected by colonoscopy biopsy for WES and customized panel design, and peripheral blood samples will be collected for baseline MRD detection ( MRD1 ) and during neoadjuvant concurrent chemoradiotherapy ( MRD2-6 ) .Peripheral blood sample will be collected 3-4 weeks after radical surgery ( MRD7 ). For patients who achieved cCR after the end of neoadjuvant therapy and adopted the W & W ( watch and wait ) strategy, the sampling time point was 3 months after the start of watching and waiting ( MRD7 ).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75
2. Rectal adenocarcinoma confirmed by pathology
3. The clinical stage is II-III.
4. Neoadjuvant chemoradiotherapy + radical surgery is planned ( cCR patients can choose to wait for observation ).
5. ECOG 0-1;
6. No distant metastasis ;
7. Main organ function is normal ;
8. signed informed consent and willing to accept long-term follow-up；
9. No anti-tumor treatment was received within 4 weeks before baseline sampling ;
10. Adequate ' colonoscopy ' tumor tissue samples can be provided for MRD customization, and sufficient whole blood samples need to be provided for baseline MRD detection.

    -

Exclusion Criteria:

1. unable to provide sufficient tissue / blood samples to meet the research needs ;
2. received radiotherapy, chemotherapy, or other targeted or immunotherapy before enrollment ;
3. Patients did not receive neoadjuvant therapy according to the original plan ;
4. Patients refused to accept genetic testing. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study intends to include 50 patients with stage II-III rectal cancer who plan to receive neoadjuvant chemoradiotherapy between the ages of 18-75 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve (AUC) of the MRD biomarker | Baseline to 12 months
  The area under the ROC curve ( AUC ) of MRD

SECONDARY OUTCOMES:
Local recurrence-free survival（LRFS） | From date of radical surgery to local recurrence or death due to disease progression，assessed up to 60 months.
  LRFS differences in patients with MRD clearance / decrease / increase
Distant metastases-free survival（DMFS） | From date of the beginning of neoadjuvant chemoradiotherapy to disease metastasis or death due to any cause,assessed up to 60 months.
  DMFS differences in patients with MRD clearance / decrease / increase

CONTACTS AND LOCATIONS:
Locations (1):
- WeiWei Xiao, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang Y, Xu H, Chen G, Pan Y. Stratified Prognostic Value of Pathological Response to Preoperative Treatment in yp II/III Rectal Cancer. Front Oncol. 2021 Dec 16;11:795137. doi: 10.3389/fonc.2021.795137. eCollection 2021. PMID 34976836
- [Background] Scholer LV, Reinert T, Orntoft MW, Kassentoft CG, Arnadottir SS, Vang S, Nordentoft I, Knudsen M, Lamy P, Andreasen D, Mortensen FV, Knudsen AR, Stribolt K, Sivesgaard K, Mouritzen P, Nielsen HJ, Laurberg S, Orntoft TF, Andersen CL. Clinical Implications of Monitoring Circulating Tumor DNA in Patients with Colorectal Cancer. Clin Cancer Res. 2017 Sep 15;23(18):5437-5445. doi: 10.1158/1078-0432.CCR-17-0510. Epub 2017 Jun 9. PMID 28600478
- [Background] Zhou J, Wang C, Lin G, Xiao Y, Jia W, Xiao G, Liu Q, Wu B, Wu A, Qiu H, Zhang F, Hu K, Xue H, Shen Z, Wang Z, Han J, Niu B, Xu Y, Yu Z, Yang L. Serial Circulating Tumor DNA in Predicting and Monitoring the Effect of Neoadjuvant Chemoradiotherapy in Patients with Rectal Cancer: A Prospective Multicenter Study. Clin Cancer Res. 2021 Jan 1;27(1):301-310. doi: 10.1158/1078-0432.CCR-20-2299. Epub 2020 Oct 12. PMID 33046514
- [Background] Pazdirek F, Minarik M, Benesova L, Halkova T, Belsanova B, Macek M, Stepanek L, Hoch J. Monitoring of Early Changes of Circulating Tumor DNA in the Plasma of Rectal Cancer Patients Receiving Neoadjuvant Concomitant Chemoradiotherapy: Evaluation for Prognosis and Prediction of Therapeutic Response. Front Oncol. 2020 Jul 24;10:1028. doi: 10.3389/fonc.2020.01028. eCollection 2020. PMID 32793464
- [Background] Wang Y, Yang L, Bao H, Fan X, Xia F, Wan J, Shen L, Guan Y, Bao H, Wu X, Xu Y, Shao Y, Sun Y, Tong T, Li X, Xu Y, Cai S, Zhu J, Zhang Z. Utility of ctDNA in predicting response to neoadjuvant chemoradiotherapy and prognosis assessment in locally advanced rectal cancer: A prospective cohort study. PLoS Med. 2021 Aug 31;18(8):e1003741. doi: 10.1371/journal.pmed.1003741. eCollection 2021 Aug. PMID 34464382